CLINICAL TRIAL: NCT00231673
Title: A Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Effect of Topiramate on Electrophysiological Parameters in Subjects With Diabetic Peripheral Polyneuropathy
Brief Title: A Study To Evaluate The Effect Of Topiramate On Clinical And Electrophysiological Parameters In Subjects With Diabetic Peripheral Polyneuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003202
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-04

CONDITIONS: Diabetic Neuropathies; Diabetes Mellitus, Type 2; Polyneuropathies
Keywords: Diabetic peripheral polyneuropathy; Electrophysiology; Nerve Conduction Study; Neurological Examination; Quantitative Sensory Testing; Topiramate
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 2; Polyneuropathies | interventions — Topiramate

ARMS (1):
- 001 (Experimental): Topiramate Increasing dosing of topiramate gradually to 200 mg daily by mouth dose maintenance for 12 weeks then decreasing dose until stopped over 12 weeks
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Increasing dosing of topiramate gradually to 200 mg daily by mouth, dose maintenance for 12 weeks, then decreasing dose until stopped over 12 weeks

SUMMARY:
The purpose of the study is to evaluate the effect of topiramate on clinical and electrophysiological parameters in patients with diabetic peripheral polyneuropathy. The study will also evaluate the safety of topiramate in this patient population.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, placebo-controlled study to evaluate the effect of topiramate on clinical and electrophysiological parameters in patients with diabetic peripheral polyneuropathy. Patients will undergo the Baseline Phase when they are tapered off other pain medications, have diabetes controlled and eligibility reassessed. Patients will then be randomized to receive either topiramate or placebo and enter the Double-Blind Phase, which consists of Titration Period (topiramate dose will be titrated from 25mg/day to 200mg/day over 42 days) and Maintenance Period (study medication will be continued for 12 weeks). After the Double-Blind Phase, study medication will be tapered off during the Taper Phase, whose duration will vary depending on each patient. The evaluations include electrophysiological assessment, quantitative sensory assessment, and clinical assessment such as subjective pain scales. Safety evaluations (vital signs, clinical laboratory evaluations, physical and neurological examination, and evaluations of adverse events) will be conducted during the trial. During the first 42 days, doses of topiramate gradually increase to achieve the target dose (200mg daily by mouth), and then the dose is maintained for 12 weeks, after which the dose is slowly reduced and stopped over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* Pain for at least 6 months prior to randomization that the investigator attributes to diabetic peripheral polyneuropathy
* Two sets of baseline nerve conduction studies and Quantitative Sensory Testing
* HbA1c =< 9%
* Diabetes controlled on stable regimen
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Diagnosis of Type 1 diabetes mellitus
* Polyneuropathy due to other underlying causes
* Hospitalization within the past 3 months due to episodes of hyper/hypoglycemia
* Other unstable medical conditions
* History of suicidal attempts
* Exposure to any other experimental drugs or device within the past 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2001-07; Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Change in peroneal nerve conduction velocity (NCV) from baseline to the end of the double-blind phase.

SECONDARY OUTCOMES:
Changes from baseline to the end of the double-blind phase in NCVs of the sural sensory nerve and ulnar (motor and sensory) nerve, and changes in amplitudes and latencies of the peroneal motor, sural sensory, and ulnar nerves. Adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study To Evaluate The Effect Of Topiramate On Clinical And Electrophysiological Parameters In Subjects With Diabetic Peripheral Polyneuropathy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=508&filename=CR003202_CSR.pdf